CLINICAL TRIAL: NCT05355428
Title: Analysing Gastric Residual Volumes in Infants Fed With Breast Milk 3 Hours Prior to General Anaesthesia
Brief Title: Reducing Fasting Time for Breast Milk to 3 Hours
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 314367
Record Dates: First submitted 2022-03-22; First posted 2022-05-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-08

CONDITIONS: Gastric Residual Volume
Keywords: anaesthesia; ultrasound; Breast milk; fasting; gastric
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- recruited patients: recruited patients will be required to feed 3 hours prior to planned procedure start with their normal method of taking breast milk (from the breast, or expressed into a bottle).
  Interventions: Other: offering of breast milk feed 3 hours prior to planned surgery start

INTERVENTIONS:
Other: offering of breast milk feed 3 hours prior to planned surgery start — parents will be asked to offer a breast milk feed (from breast or expressed in bottle) at a given time 3 hours prior to planned induction time

SUMMARY:
Shortening fasting times in young children undergoing general anesthesia aims to avoid the detrimental effects of prolonged fasting. However, the quantities of acidified milk that might be expected in the stomach following a shortened fast have not yet been fully investigated. The role of gastric ultrasound in quantifying particulate gastric content is not fully understood.

DETAILED DESCRIPTION:
Prolonged fasting prior to general anaesthesia (GA) is common in children. It is associated with dehydration, hypoglycemia, and ketoacidosis in up to 28 % of children under 3 years, as well as distress in children and their families.

The purpose of pre-operative fasting is to reduce the volume, acidity, and particulate nature of any gastric contents; therefore, if an aspiration event occurs, lung damage will be minimal. Although pulmonary aspiration events are rare in children, data from animal models suggest that the volume, and presence of particulate matter, such as that seen in acidified breast or formula milk, can affect the patterns of lung damage. Aspiration of volumes greater than 0.8 ml.kg-1 appear to be the most harmful in animal models, regardless of pH.

In humans, gastric emptying of breast and formula milk preparations has been extensively studied in the neonatal setting in preterm and low-birth-weight infants. The majority used serial measurements of antral cross-sectional area (ACSA) with gastric ultrasound (US) and reported the return of ACSA values to baseline within 3 h for breast milk and 4 h for formula milk.

The European Society of Anesthesia and Intensive Care published guidance in 2022, advocating a 3-hour breast milk fast, and a 4-hour formula milk fast in children under 1 year undergoing elective GA. This guidance has been adopted in some tertiary centers in the UK despite the paucity of prospective studies investigating the impact of a shortened fast on gastric residual volume (GRV) measured directly (for example, by gastric aspiration).

In 2011, using data from adult elective surgical patients, Perlas et al. devised a qualitative assessment grading system to assess the gastric antrum prior to induction [15], with a view to guiding decision making regarding the induction method. various formulae that incorporate antrum grade and antrum cross sectional area have subsequently been devised and validated in adults and children over 1 year of age.

A formula devised by Kim et al. demonstrated good correlation with suctioned gastric volumes in anesthetized children under 1 year of age. It is not known whether a formula derived from data in a cohort of children with clear fluid gastric content resulting from a prolonged overnight fast will perform as well in a cohort of young children who have recently been fed, where, if present, gastric content may be semi-solid or particulate.

The primary aims of this study were to measure GRV of gastric contents measured by naso-gastric aspiration in infants who were breast fed 3 hours prior to general anesthesia. The secondary aim is to correlate predicted GRV using a mathematical formula proposed by Kim et al, to measure GRV by NG aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Babies born at or after 37 weeks post menstrual age
* Babies born prior to 37 weeks who are now more than 37 weeks corrected post menstrual age (PMA)
* Elective surgery
* Breast fed including expressed breast milk, in isolation or combination with solids or formula.

Exclusion Criteria:

* Babies who are less than 37 weeks PMA,
* Ex-premature babies who are now greater than 37 weeks PMA but who have significant lung, heart, kidney or liver disease.
* Known delayed gastric emptying

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Breast fed children under 18 months of age, presenting for elective procedures under general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Gastric residual volume | 12 months
  Ascertain the residual volume of gastric contents in 50 infants who are given breast milk 3 hours prior to general anaesthesia

SECONDARY OUTCOMES:
Gastric ultrasound | 12 months
  The secondary aim of this study is to ascertain how well ultrasound derived measurement of gastric residual volume correlates to direct measurement via nasogastric tube aspiration.

CONTACTS AND LOCATIONS:
Locations (1):
- Emily Saffer, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
On reasonable request data can be supplied

REFERENCES:
- [Background] Perrella SL, Hepworth AR, Gridneva Z, Simmer KN, Hartmann PE, Geddes DT. Gastric Emptying and Curding of Pasteurized Donor Human Milk and Mother's Own Milk in Preterm Infants. J Pediatr Gastroenterol Nutr. 2015 Jul;61(1):125-9. doi: 10.1097/MPG.0000000000000776. PMID 25729886
- [Result] Litman RS, Wu CL, Quinlivan JK. Gastric volume and pH in infants fed clear liquids and breast milk prior to surgery. Anesth Analg. 1994 Sep;79(3):482-5. doi: 10.1213/00000539-199409000-00013. PMID 8067551
- [Result] van der Walt JH, Foate JA, Murrell D, Jacob R, Bentley M. A study of preoperative fasting in infants aged less than three months. Anaesth Intensive Care. 1990 Nov;18(4):527-31. doi: 10.1177/0310057X9001800420. PMID 2268020
- [Result] Walker RW. Pulmonary aspiration in pediatric anesthetic practice in the UK: a prospective survey of specialist pediatric centers over a one-year period. Paediatr Anaesth. 2013 Aug;23(8):702-11. doi: 10.1111/pan.12207. Epub 2013 Jun 13. PMID 23763657
- [Result] Warner MA, Warner ME, Warner DO, Warner LO, Warner EJ. Perioperative pulmonary aspiration in infants and children. Anesthesiology. 1999 Jan;90(1):66-71. doi: 10.1097/00000542-199901000-00011. PMID 9915314
- [Result] Tan Z, Lee SY. Pulmonary aspiration under GA: a 13-year audit in a tertiary pediatric unit. Paediatr Anaesth. 2016 May;26(5):547-52. doi: 10.1111/pan.12877. Epub 2016 Mar 17. PMID 26990683
- [Result] Ewer AK, Yu VY. Gastric emptying in pre-term infants: the effect of breast milk fortifier. Acta Paediatr. 1996 Sep;85(9):1112-5. doi: 10.1111/j.1651-2227.1996.tb14227.x. PMID 8888928
- [Result] MASON S. Some aspects of gastric function in the newborn. Arch Dis Child. 1962 Aug;37(194):387-91. doi: 10.1136/adc.37.194.387. No abstract available. PMID 14470855
- [Result] Van Den Driessche M, Peeters K, Marien P, Ghoos Y, Devlieger H, Veereman-Wauters G. Gastric emptying in formula-fed and breast-fed infants measured with the 13C-octanoic acid breath test. J Pediatr Gastroenterol Nutr. 1999 Jul;29(1):46-51. doi: 10.1097/00005176-199907000-00013. PMID 10400103
- [Result] Cavell B. Gastric emptying in infants fed human milk or infant formula. Acta Paediatr Scand. 1981 Sep;70(5):639-41. PMID 7324911
- [Result] Beck CE, Witt L, Albrecht L, Winstroth AM, Lange M, Dennhardt N, Boethig D, Sumpelmann R. Ultrasound assessment of gastric emptying time in preterm infants: A prospective observational study. Eur J Anaesthesiol. 2019 Jun;36(6):406-410. doi: 10.1097/EJA.0000000000001007. PMID 31021881
- [Result] Italianer MF, Naninck EFG, Roelants JA, van der Horst GTJ, Reiss IKM, Goudoever JBV, Joosten KFM, Chaves I, Vermeulen MJ. Circadian Variation in Human Milk Composition, a Systematic Review. Nutrients. 2020 Aug 4;12(8):2328. doi: 10.3390/nu12082328. PMID 32759654
- [Result] Kent JC, Mitoulas LR, Cregan MD, Ramsay DT, Doherty DA, Hartmann PE. Volume and frequency of breastfeedings and fat content of breast milk throughout the day. Pediatrics. 2006 Mar;117(3):e387-95. doi: 10.1542/peds.2005-1417. PMID 16510619
- [Result] Janahi IA, Elidemir O, Shardonofsky FR, Abu-Hassan MN, Fan LL, Larsen GL, Blackburn MR, Colasurdo GN. Recurrent milk aspiration produces changes in airway mechanics, lung eosinophilia, and goblet cell hyperplasia in a murine model. Pediatr Res. 2000 Dec;48(6):776-81. doi: 10.1203/00006450-200012000-00013. PMID 11102546
- [Result] O'Hare B, Chin C, Lerman J, Endo J. Acute lung injury after instillation of human breast milk into rabbits' lungs: effects of pH and gastric juice. Anesthesiology. 1999 Apr;90(4):1112-8. doi: 10.1097/00000542-199904000-00026. PMID 10201684
- [Result] Yigit S, Akgoz A, Memisoglu A, Akata D, Ziegler EE. Breast milk fortification: effect on gastric emptying. J Matern Fetal Neonatal Med. 2008 Nov;21(11):843-6. doi: 10.1080/14767050802287176. PMID 18985557
- See also: Gastric Emptying and Intragastric Behavior of Breast Milk and Infant Formula in Lactating Mothers — https://doi.org/10.1093/jn/nxab295

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT05355428/Prot_SAP_000.pdf